CLINICAL TRIAL: NCT05354882
Title: Interventional Study on DEterminants and Factors of Physical ACtivity After Treatments in Oncology
Acronym: DEFACTO2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Sorbonne Paris Nord (Other)
Collaborators: Ligue contre le cancer, France (Other); Garmin International (Industry); Stimulab (Unknown)
Responsible Party: Principal Investigator, Audemarie Foucaut, Associate Professor, Université Sorbonne Paris Nord
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-A01570-41
Record Dates: First submitted 2022-04-11; First posted 2022-05-02 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Colo-rectal Cancer; Lung Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms; Prostatic Neoplasms | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Feasibility group. Single group (intervention group) will be given access to the DEFACTO intervention for twelve-weeks.
  Interventions: Behavioral: Physical activity program

INTERVENTIONS:
Behavioral: Physical activity program — The single group will access to the twelve-week DEFACTO program containing one adapted physical activity session, two discussion group sessions and several motivational interviewing
  Other Names: Motivational Interviewing; Discussion group; Adapted physical activity

SUMMARY:
Benefits of physical activity (PA) as supportive care in cancer have been widely demonstrated by the scientific community. However, survivors who have completed chemo-radio-immunotherapy treatments doesn't achieve PA recommendations on average. This reinforces the need to identify factors influencing PA level, and to propose a multilevel model (macro-, meso-, micro-level) to understand better what facilitates the adoption and maintenance of active behaviour and what hinders it. To date, there is no ecological model in France explaining this behaviour in the post-treatment phase of breast, colorectal, prostate, and lung cancers. From this initial model, we seek to design an educational and motivational intervention in PA.

Thus, the investigators propose to test the feasibility of implementing an individualized program to increase and maintain level of physical activity and to decrease sedentary behaviours in physically inactive cancer survivors. This program is based through and identification of barriers and facilitators of an active lifestyle among this population.

DETAILED DESCRIPTION:
In 2008, 3 million French people had experienced cancer in the last 15 years, compared to 18 million in 2022. Post-treatment marks a break with the intensive care pathway. It frequently leads to changes in the lifestyle of these patients. During this period, behaviors conducive to maintaining their state of health remain important.

Among these behaviors, Physical Activity (PA) is an integral part and brings many post-treatment benefits. Despite the evidence of PA benefits in adult cancer survivors who have completed chemo-radio-immunotherapy treatments, the majority of those with good prognosis cancer are insufficiently active. Patient survival tends to increase by 20% thanks to scientific progress and the improvement of cancer management. At the same time, patients experience adverse effects for an extended period after cancer treatment. It would take an average of 10 to 15 years to note a decrease in the psychological, physical, professional, and socio-economic repercussions of cancer. These repercussions do not totally disappear over time. We have a particular interest in this post-treatment period, where the end of treatments marks a break within the "clinical pathway". The patient then joins the "care pathway" where he/she needs to have an autonomous management of his/her health behaviour.

The study of factors - clinical, psychological, cognitive, behavioural, social, or even linked to the clinical pathway and the geographical environment - involved in regular PA practice with breast, prostate, colorectal, or lung cancer survivors, would allow us an overview of what shapes a complex behaviour like PA.

In view of these needs to better understand and act on the complex behaviour of active lifestyle, the main objective of our research is to design, implement, and evaluate an individualised educational and motivational program, constructed from an explanatory ecological model. The educational and motivational program thus conceived will help in supporting good prognosis and physically inactive cancer survivors (breast, colorectal, prostate, or lung cancers) in initiation and maintenance of their PA.

Deployment of this interventional approach will provide more support to cancer survivors at the end of their treatment at a national level while considering the specificities of healthcare fields. To consider these variety, transferability criteria will be taken into account.

Thus, the investigators propose to test the feasibility of implementing an individualized program to increase and maintain level of physical activity and to decrease sedentary behaviours in physically inactive cancer survivors. This program is based through and identification of barriers and facilitators of an active lifestyle among this population.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ age < 75 years
* survivors of primary non-metastatic breast, lung, prostate or colorectal cancer (stage I, II or III and primary, second and relapse included)
* 3 weeks to 20 years post-treatment (surgery, chemotherapy, radiation therapy and/or immunotherapy) not including hormonal therapy
* Whose ability to participate in the APA intervention has been certified by a medical certificate issued by physician
* Availability and willingness to invest in the DEFACTO study during the program (3 months) and during the post-program follow-up (12 months)
* Participating, on average, in no more than 150 minutes of moderate physical activity or no more than 75 minutes of vigorous activity per week
* Average at least 6 hours a day of sedentary behaviours
* Able to read, understand and complete questionnaires in French
* Able to use connected device (Vivosmart4®) and to perform simple operating actions (press a button, recharge the battery)
* possessing a smartphone which can download Garmin Connect application ®
* Able to walk unassisted
* French speaking and living in France
* having signed the consent form

Exclusion Criteria:

* Current evidence of metastatic disease
* Having an absolute contraindication by a physician to practice PA
* Using treatments that influence blood pressure, cardiotoxic drugs, painkillers (morphinics);
* Using cane or walking aid
* Deprived of liberty by judicial or administrative decision
* Person under guardianship or curatorship
* Pregnancy and/or lactating women
* Being diagnosed of any cardiac abnormalities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change of physical activity (connected device) | One week before initiation of DEFACTO intervention, during the intervention and intervention at Month 3 and Month 6 and Month 12
  Average daily steps, distance traveled, floors climbed, heart rate, cumulative duration of activities of moderate and vigorous intensities using VIVOSMART4® (Garmin)

SECONDARY OUTCOMES:
Change of physical activity by the Global Physical Activity Questionnaire (GPAQ) | At baseline (at inclusion), and at the completion of intervention (12 weekends after the start of the intervention)
  Change of physical activity evaluated by the GPAQ questionnaire, at baseline (at inclusion), and at the completion of intervention (12 weekends after the start of the intervention)
Assessment of life quality | At Baseline (at inclusion), and at the completion of intervention (12 weekends after the start of the intervention)
  Assessment by using the Short-Form 12 questionnaire (SF-12) Life quality scores calculation
Assessment of Health literacy level | At Baseline (at inclusion), and at the completion of intervention (12 weekends after the start of the intervention)
  Assessment by using a single question concerning the need to resort refer to a health professional to understand health information
Assessment of Knowledge about PA and its link with cancer | At Baseline (at inclusion), and at the completion of intervention (12 weekends after the start of the intervention)
  Assessment by using specific questions of the Cancer Exercise Stereotypes Scale
Physical activity barriers | At Baseline (at inclusion), and at the completion of intervention (12 weekends after the start of the intervention)
  Assessment by using the "General determinants of PA" questionnaire. This tool examines 7 areas: 1) Lack of time; 2) Social influences; 3) Lack of energy; 4) Lack of willingness; 5) Fear of hurting yourself; 6) Lack of skill sets; 7) Lack of resources
Transtheorical model's variables related to physical activity | At Baseline (at inclusion), and at the completion of intervention (12 weekends after the start of the intervention)
  Assessment by using the "Stages of change" questionnaire, "Processes of change (POC)" questionnaire, "decisional balance" questionnaire, and "self-efficacy" questionnaire.
Motivation to physical activity pratice | At Baseline (at inclusion), and at the completion of intervention (12 weekends after the start of the intervention)
  Types of motivation based on self-determination theory, assessment by using the Motivation Scale for by Physical Activity for Health Purposes

OTHER OUTCOMES:
Weight | At Baseline (at inclusion)
  in kilograms (weight and height will be combined to report BMI in kg/m^2)
Height | At Baseline (at inclusion)
  in centimeters (height and weight will be combined to report BMI in kg/m^2)
Date of cancer diagnosis | At Baseline (at inclusion)
  (month/year)
Tumor location and cancer recurrence or second primary cancer | At Baseline (at inclusion)
  (breast, colorectal, lung or prostate)
Stage of cancer | At Baseline (at inclusion)
  (I, /II, or /III)
Type of treatment | At Baseline (at inclusion)
  (chemotherapy, radiation therapy, immunotherapy, hormonotherapy)
Clinical data | At Baseline (at inclusion)
  Body Mass Index (BMI, kg/m^2), date of diagnosis (month/year), tumour location (breast, colorectal, lung or prostate), stage of cancer (I, /II, or /III), cancer recurrence or second primary cancer, type of treatment, date on the treatment end (chemotherapy, radiation therapy, immunotherapy, hormonotherapy + month/year); (close-ended questions)
Date on the treatment end | At Baseline (at inclusion)
  (month/year)
Socio-demographic variables | At Baseline (at inclusion)
  Educational qualifications, economic class-status, current professional situation, household type, habitat type, geographical environment (rural or /urban); (close-ended questions)

CONTACTS AND LOCATIONS:
Overall Officials: Aude-Marie AF Foucaut, Principal Investigator — Université Sorbonne Paris Nord, Laboratoire Educations et Promotion de la Santé UR3412
Locations (1):
- Laboratoire Educations et Promotion de la Santé UR3412, Bobigny, France

REFERENCES:
- [Derived] Aumaitre A, Gagnayre R, Foucaut AM. Determinants and Factors of Physical Activity After Oncology Treatments (DEFACTO) in Metropolitan France: Protocol of a Mixed Methods Study and Intervention. JMIR Res Protoc. 2024 May 16;13:e52274. doi: 10.2196/52274. PMID 38753415

DOCUMENTS (1):
  • Informed Consent Form (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT05354882/ICF_000.pdf